CLINICAL TRIAL: NCT07358949
Title: Feasibility and Acceptability of Point of Care Rapid Syphilis Testing Among Patients Seeking Family Planning Services in Hawai'i
Status: Not yet recruiting | Type: Observational
Sponsor: Queen's Medical Center (Other)
Responsible Party: Principal Investigator, Elaine Chan, Complex Family Planning Fellow, Queen's Medical Center
Other Study IDs: RA-2026-xxx
Record Dates: First submitted 2025-12-31; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Syphilis Infection
Keywords: feasibility; rapid syphilis testing; family planning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid Syphilis Test — This study aims to evaluate whether the Syphilis Health Check (SHC), an FDA-approved rapid, point-of-care syphilis test, is feasible and acceptable to patients and providers at a university-associated family planning clinic in Hawai'i.
  SHC is specific for detecting Treponema pallidum antibodies in serum, plasma, or whole blood via a rapid immunochromatographic test. It has a sensitivity of 95-99% and a specificity of 94-97%, and has been studied in pregnant patients. The test costs approximately $10, takes 10-15 minutes to yield results, has a shelf life of 30 months, and remains stable at room temperature. The assay can be used as an initial screening test or in conjunction with a non-treponemal laboratory test. Treatment with antibiotics can be started immediately with a positive SHC test.

SUMMARY:
The purpose of the study is to see if rapid syphilis testing at the time of a family planning (contraception or abortion) visit is acceptable and practical for patients.

This study involves a fingerstick blood sample for syphilis testing during a family planning visit. Results will be ready in 10-15 minutes.

Potential Benefits

* Participants can find out whether they are syphilis positive or negative within the visit, as soon as 10-15 minutes of the finger stick. Typically, syphilis testing results take several days.
* If positive, there is the option of starting treatment within the same day.

Potential Risks

* The study team will do everything possible to protect participants' privacy, including removing names and other identifiable information from study materials, however this is still a small chance there may be a breach of privacy during the study.
* Physical risks of fingerstick are exceptionally rare when sterile technique is used. The study team will be using all best practices to reduce risk of infection or injury.
* There is a risk of discomfort or pain with fingerstick collection. The risk of scarring is usually only associated with repeat draws, for example in patients with diabetes who have to do fingerstick draws multiple times per day.
* There is a very small chance that the positive result is incorrect (also known as a "false positive"), meaning the participant does not actually have syphilis. To confirm the result, the investigators recommend that any positive rapid syphilis result be followed up with a blood test at the lab.

Cost for Participation

o There is no cost to participate in this study. If the participant tests positive for syphilis, the study will help cover the cost of treatment if not continuing the pregnancy. If the participant chooses to continue the pregnancy, the study team will refer the participant to the Department of Health for management of treatment. The participant or their insurance may be responsible for costs associated with treatment in this scenario.

DETAILED DESCRIPTION:
This is a nonrandomized feasibility study of a clinician-administered point of care rapid syphilis test. The study will take place within the Queen's Medical Center Options Clinic, where the University of Hawai'i Complex Family Planning program is based. The Options Center is a primary referral site for abortion throughout Hawai'i. This study aims to evaluate whether the Syphilis Health Check (SHC), an FDA-approved rapid, point-of-care syphilis test, is feasible and acceptable to patients and providers at a university-associated family planning clinic in Hawai'i. Rapid syphilis testing will be offered to sexually active adults seeking abortion or contraception services. Positive results will be followed by laboratory-based syphilis testing. The investigators hypothesize that rapid syphilis testing at the family planning clinic will be feasible and acceptable to both patients and staff.

If the patient expresses interest in syphilis testing, a research associate will describe the study in further detail and obtain informed consent via a paper-based informed consent document.

All study personnel will undergo the SHC training, which includes an online module and quiz available on the SHC website. Study personnel who are certified to collect the SHC will collect the specimen via fingerstick using a sterile lancet. They will collect the blood using the pipette provided in each kit, then add the blood to the sample well of the SHC cassette. They will then add four drops of diluent to the sample well. The study personnel can read the result at the 10-minute mark, and no later than 15 minutes. Any line in the 'T' zone, even if faint, accompanied by a line in the 'C' zone, will be interpreted as a positive result. The study personnel, if not a family planning provider, will inform the physician of all test results. All participants with a positive SHC test will be recommended to get confirmatory serological testing. All participants will receive their results before the end of their family planning visit.

Traditional serological testing requires external laboratory equipment and facilities. The SHC is read in the clinic without additional equipment or laboratory technicians, thus expediting time from specimen collection to diagnosis. Participants with positive SHC results will require more thorough evaluation to stage and determine appropriate treatment. The physician will conduct a detailed health history and physical exam. The SHC is a qualitative treponemal test; therefore, after their counseling and discussion with the physician, the participant will be asked to go to the laboratory to draw blood for an RPR, for which there is no rapid test. The RPR acts as a confirmatory test while also providing quantitative information to monitor treatment effectiveness.

If the participant is pregnant and desires to continue with pregnancy, then the patient will be referred to a pharmacy or clinic that can administer Bicillin. These may include Queen's pharmacy, other pharmacy, Healthy Mothers Healthy Babies, PATH Clinic, Diamond Head STI Clinic. Additional appointments as needed will be made to complete the treatment (up to 3 total doses of Bicillin). If there is still an ongoing shortage and/or recall of Bicillin at the time of study initiation, the physician will call 808-833-9281 to request an appointment with the Hawai'i Department of Public Health STI/HIV Clinic for assistance with where to refer the patient for Bicillin treatment options. At the time of writing, Bicillin is prioritized for pregnant individuals only. For participants with positive SHC who are terminating pregnancy or who are not pregnant, the alternative treatment is doxycycline per CDC guidelines. The physician will prescribe 2 to 4 weeks of doxycycline 100mg BID based on the staging of infection in accordance with CDC guidelines. Patients will be counseled on increased sun sensitivity with longer durations of doxycycline use, and recommend sun protection.

Positive SHC results that have been confirmed with positive serum RPR will be reported to the State of Hawai'i Department of Health using the Sexually Transmitted Infection Confidential Case Report within three business days per state guidelines, either through mail, fax, or phone .

For partner notification, the study physician will provide resources for patients to share with their partner(s) for testing options. Options will include: 1) the patient informs their sexual partner(s) directly or anonymously through a text-based service; 2) the physician informs their sexual partner(s) via a text-based service; 3) deferring to the public health department to inform their sexual partner(s) through their intervention specialist team.

ELIGIBILITY:
Inclusion Criteria:

* 14 years or older
* Seeking contraception or abortion services
* Sexually active (engages in any form of sexual activity with another person)
* Denies history of syphilis infection
* Can speak and read English
* Displays capacity for informed consent

Exclusion Criteria:

* Confirmed history (by patient report or medical records) of syphilis
* Home address outside Hawai'i
* Currently incarcerated

Number of Subjects:

Recommendations for sample size in pilot studies range from 70 to 100 patients.28 Given this is a nonrandomized feasibility study with no comparator (i.e., to a control or to serological testing), we aim to enroll 50 to 75 participants to support analysis for correlation between variables while being able to achieve relatively small confidence intervals. This number takes into account the practical considerations of study personnel resources and in-person patient volume in our clinic. All patients eligible for the rapid syphilis testing will be approached for study participation.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Queens Options Center serves as a referral center for family planning services for patients throughout the state. From prior literature, the patients most impacted by persistent or continued syphilis infections are those who are structurally vulnerable, including those who are under- or uninsured, experiencing poverty, unhoused, or actively using substances. By screening universally, we may decrease the stigmatization associated with individual behavior-based screening. We acknowledge that there is a risk of increased false positives by screening universally . To mitigate this, we recommend that a participant with a positive rapid test also obtain serological testing with RPR, which is already required for treatment monitoring. As stated above, prior studies have established that the sensitivity and specificity of the SHC are greater than 95%.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability and Feasibility of Rapid Syphilis Testing | 12 months
  We will assess feasibility with a combination of quantitative and qualitative methods, in accordance with guidelines put forth by Teresi et al for feasibility pilot studies.
  Outcomes:
  * Number of eligible participants
  * Number of participants who completed SHC testing
  * Number of participants who agreed to SHC testing
  * Number of participants able to obtain SHC result
  * To calculate feasibility, the proportion of all eligible patients who completed testing will be determined.
  * To calculate completion rate of the SHC tests using the number of participants who were able to obtain an SHC result divided by the number of participants who agreed to rapid syphilis testing.
  Descriptive statistics will be used to assess acceptibility.

SECONDARY OUTCOMES:
Secondary Outcomes | 12 months
  Secondary outcomes:
  * Number of family planning patients who had syphilis testing in the past year.
  * Number of family planning patients who test positive for syphilis.
  * Time (in days) to prescribe treatment after positive syphilis test.
Assess the acceptability and feasibility of a point-of-care rapid syphilis testing in a university-affiliated family planning clinic. | 12 months
  We will assess feasibility with a combination of quantitative and qualitative methods, in accordance with guidelines put forth by Teresi et al for feasibility pilot studies.
  Outcomes:
  * Number of eligible participants
  * Number of participants who completed SHC testing
  * Number of participants who agreed to SHC testing
  * Number of participants able to obtain SHC result
  * To calculate feasibility, the proportion of all eligible patients who completed testing will be determined.
  * To calculate completion rate of the SHC tests using the number of participants who were able to obtain an SHC result divided by the number of participants who agreed to rapid syphilis testing.
  * Descriptive statistics will be used to assess acceptibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Medical Center, 1004 Clinic POB1, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Result] Harvey L, Jacka B, Bazerman L, Thomas A, Moody M, Irvin R, Beckwith CG. Feasibility and Performance of a Point-of-Care Hepatitis C RNA Assay in a Community Supervision Cohort. JAMA Netw Open. 2024 Oct 1;7(10):e2438222. doi: 10.1001/jamanetworkopen.2024.38222. PMID 39374019
- [Result] Nuwagaba-Biribonwoha H, Simelane S, Sithole T, Dlamini S, Mavimbela M, Dube N, Mamba S, Mamba M, Sahabo R, El Sadr WM, Abrams EJ, Justman J. Feasibility and Acceptability of Point-of-Care Testing for Sexually Transmitted Infections in Outpatient Clinics Offering Integrated Services in Eswatini. Sex Transm Dis. 2024 Nov 1;51(11):743-749. doi: 10.1097/OLQ.0000000000001997. Epub 2024 Jun 11. PMID 38860665
- [Result] Stafford I, Bakunas C, Haydamous J, Mosqueda A, Klausner JD, Mena L, Blackwell SC. Implementation of an Opt-Out and Rapid Point-of-Care Syphilis Testing Program for Pregnant Patients Presenting to the Emergency Department. Sex Transm Dis. 2025 Jun 1;52(6):352-355. doi: 10.1097/OLQ.0000000000002131. Epub 2024 Dec 24. PMID 39718531
- [Result] Missed Opportunities for Prevention of Congenital Syphilis -United States, 2018. Pediatr Infect Dis J. 2020 Nov 1;39(11):1062. doi: 10.1097/INF.0000000000002833. No abstract available. PMID 33369594
- [Result] Corrigendum to "Syphilis Screening: A Review of the Syphilis Health Check Rapid Immunochromatographic Test". J Pharm Technol. 2020 Apr;36(2):91. doi: 10.1177/8755122520904797. Epub 2020 Jan 29. PMID 34752533
- [Result] Cao W, Thorpe PG, O'Callaghan K, Kersh EN. Advantages and limitations of current diagnostic laboratory approaches in syphilis and congenital syphilis. Expert Rev Anti Infect Ther. 2023 Jul-Dec;21(12):1339-1354. doi: 10.1080/14787210.2023.2280214. Epub 2023 Nov 24. PMID 37934903
- [Result] Chan EYL, Smullin C, Clavijo S, Papp-Green M, Park E, Nelson M, Giarratano G, Wagman JA. A qualitative assessment of structural barriers to prenatal care and congenital syphilis prevention in Kern County, California. PLoS One. 2021 Apr 1;16(4):e0249419. doi: 10.1371/journal.pone.0249419. eCollection 2021. PMID 33793630
- [Result] Plotzker RE, Burghardt NO, Murphy RD, McLean R, Jacobson K, Tang EC, Seidman D. Congenital syphilis prevention in the context of methamphetamine use and homelessness. Am J Addict. 2022 May;31(3):210-218. doi: 10.1111/ajad.13265. Epub 2022 Mar 27. PMID 35340101
- [Result] McNicholas C, Madden T, Secura G, Peipert JF. The contraceptive CHOICE project round up: what we did and what we learned. Clin Obstet Gynecol. 2014 Dec;57(4):635-43. doi: 10.1097/GRF.0000000000000070. PMID 25286295
- [Result] Adimora AA, Schoenbach VJ. Social context, sexual networks, and racial disparities in rates of sexually transmitted infections. J Infect Dis. 2005 Feb 1;191 Suppl 1:S115-22. doi: 10.1086/425280. PMID 15627221
- [Result] Johnson KA, Snyder RE, Tang EC, de Guzman NS, Plotzker RE, Murphy R, Jacobson K. Geospatial Social Determinants of Health Correlate with Disparities in Syphilis and Congenital Syphilis Cases in California. Pathogens. 2022 May 6;11(5):547. doi: 10.3390/pathogens11050547. PMID 35631068
- [Result] Gan A, Shintaku KM, Begue RE. Gaps in the Care of Maternal and Congenital Syphilis in Hawai'i, 2022-2023. Pediatr Infect Dis J. 2025 Dec 1;44(12):e440-e445. doi: 10.1097/INF.0000000000004931. Epub 2025 Aug 6. PMID 40829011